CLINICAL TRIAL: NCT01926262
Title: Physical Exercise Against Neck and Shoulder Pain in Danish Military Helicopter Pilots and Crewmembers - A Clinical Randomized, Controlled Trail
Brief Title: Exercise as Treatment of Neck Pain Among Helicopter Pilots and Crew Members
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: The Royal Danish Air Force (Unknown)
Responsible Party: Principal Investigator, Mike Murray, MSc, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: S-20120121
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Neck Pain; Shoulder Pain
Keywords: Pain, Neck, Exercise, Pilots, Crewmembers,
MeSH Terms: conditions — Neck Pain; Shoulder Pain; Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Exercise Group (Experimental): Specific Strength Training for the Neck and Shoulder muscles
  Interventions: Behavioral: Specific Strength Training
- Reference group (No Intervention): No Specific Strength Training

INTERVENTIONS:
Behavioral: Specific Strength Training — Specific Strength Training for the Neck and Shoulder Muscles
  Arms: Physical Exercise Group

SUMMARY:
The aim of this project is to investigate, whether physical training, targeted neck and shoulder muscles, can reduce and prevent neck pain among military helicopter pilots and crewmembers.

DETAILED DESCRIPTION:
Military helicopter pilots and crewmembers is often burdened by work-related neck and shoulder pain. Neck pain is a health challenge, that can reduce functional level, concentration and operational safety. Physical exercise has shown good efficacy in reducing neck/shoulder pain in other occupational groups in previous studies.

The Royal Danish Air Force and the University of Southern Denmark, wishes to examine whether specific physical exercise can prevent and reduce neck/shoulder pain within this occupational group.

Participants in this project will be randomly selected to either a physical exercise group or a reference group.

* The physical exercise group will follow a training program targeted neck and shoulder muscles and train 1 hour per week (3 x 20 min) for 26 weeks.
* The reference group will continue normal routines, including workout routines. They will later be offered the same training program as the Physical Exercise group provided that training has a positive effect.

ELIGIBILITY:
Inclusion Criteria:

* Employed within the Royal Danish Air Force
* Helicopter pilot
* Crewmember (Flight engineer, Rescue swimmer or Mission System Operator)
* Flown within the past 6 months

Exclusion Criteria:

* Grounded at time of inclusion
* Participated in a training intervention within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Neck and shoulder pain | 6 months
  Neck pain will be assessed as self-rated pain on a 10 point scale by questionnaire at baseline and follow-up after 6 months

SECONDARY OUTCOMES:
Pressure-Pain-Threshold | 6 months
  Pressure-Pain-Threshold will be assessed at baseline and follow-up after 6 months
Muscle strength and steadiness | 6 months
  Muscle strength and steadiness will be quantified by force transducers at baseline and follow-up after 6 months
Postural stability | 6 months
  Postural stability will be assessed at baseline and follow-up after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Sjøgaard, Professor.,, Study Director — University of Southern Denmark
Locations (1):
- Hilicopter Wing Karup, Karup, Denmark

REFERENCES:
- [Derived] Murray M, Lange B, Nornberg BR, Sogaard K, Sjogaard G. Self-administered physical exercise training as treatment of neck and shoulder pain among military helicopter pilots and crew: a randomized controlled trial. BMC Musculoskelet Disord. 2017 Apr 7;18(1):147. doi: 10.1186/s12891-017-1507-3. PMID 28388892
- [Derived] Murray M, Lange B, Nornberg BR, Sogaard K, Sjogaard G. Specific exercise training for reducing neck and shoulder pain among military helicopter pilots and crew members: a randomized controlled trial protocol. BMC Musculoskelet Disord. 2015 Aug 19;16:198. doi: 10.1186/s12891-015-0655-6. PMID 26286707
- See also: University of Southern Denmark — http://www.sdu.dk/en/om_sdu/institutter_centre/iob_idraet_og_biomekanik/forskning/forskningsenheder/fysiskaktivitetsundhed